CLINICAL TRIAL: NCT02219347
Title: Biomarkers of Remission in Rheumatoid Arthritis (BioRRA)
Acronym: BioRRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Newcastle University (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NUTH7100
Record Dates: First submitted 2014-08-15; First posted 2014-08-18 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; biological markers; remission; ultrasonography; microarray; survival analysis; T cell
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DMARD cessation (Other): All patients recruited to the study who have a Disease Activity in 28 Joints C-Reactive Protein (DAS28-CRP) score of < 2.4 and who do not have power Doppler synovitis on a 7-joint musculoskeletal ultrasound scan will stop their DMARD therapy. These patients will then be followed-up for a period of 6 months or until flare of their arthritis activity, whichever is sooner.
  Interventions: Drug: DMARD cessation

INTERVENTIONS:
Drug: DMARD cessation — Complete cessation of non-biologic DMARD therapy (single or combination of methotrexate, sulphasalazine and/or hydroxychloroquine)

SUMMARY:
Rheumatoid arthritis is a common condition affecting approximately 1% of the United Kingdom population; it is an autoimmune disease where the body's natural defences (the immune system) attack the body itself resulting, most notably, in joint damage and arthritis. To help prevent this, patients with rheumatoid arthritis need to take disease-modifying anti-rheumatic drugs (DMARDs). As rheumatoid arthritis is a life-long condition, these drug treatments are prescribed as long-term medications taken for many years.

With successful drug treatment, many patients are able to achieve an excellent control of their disease and their arthritis can go in to remission. At present, there are no markers which can reliably predict which of these patients can reduce their drug treatment, and hence benefit from a lower risk of side effects and inconvenience, without an increase in their arthritis activity.

We invite patients with stable rheumatoid arthritis to participate in this study conducted by Newcastle upon Tyne Hospitals NHS Foundation Trust in collaboration with Newcastle University and funded by the Wellcome Trust. Patients whose arthritis is confirmed as being in remission will be able to stop their DMARD medication and be monitored for a period of 6 months. Patients whose arthritis activity increases during this time will be able to restart their DMARD medication, whereas those patients whose arthritis remains in remission will be able to stay off DMARD medication.

The main aim of this study is to identify clinical, ultrasound and blood markers that can predict which patients will remain in remission after stopping DMARD medication. If identified, these markers could be a useful guide to doctors and patients in the future when deciding whether to stop DMARD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rheumatoid arthritis made by consultant rheumatologist at least 12 months previously
* Current single or combination use of methotrexate, sulphasalazine and/or hydroxychloroquine
* Arthritis currently in remission, as judged clinically by referring healthcare professional
* Willing to consider DMARD withdrawal

Exclusion Criteria:

* Use of biologic therapy within the past 6 months
* Received steroids within past 3 months (enteral, parenteral or intra-articular)
* Use of any DMARD other than methotrexate, sulphasalazine or hydroxychloroquine within the past 6 months (or past 12 months for leflunomide)
* Current pregnancy, or pregnancy planned within next 6 months
* Current participation within another clinical trial
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Time-to-flare of arthritis activity following DMARD cessation | From recruitment, assessed up to 6 months
  Flare of arthritis activity defined as Disease Activity Score in 28 Joints C-Reactive Protein (DAS28-CRP) score greater than or equal to 2.4

SECONDARY OUTCOMES:
Clinical biomarkers predictive of DMARD-free remission | At recruitment
  Baseline clinical factors predictive of time-to-flare of arthritis activity following DMARD cessation.
Ultrasound biomarkers of DMARD-free remission | At recruitment
  Baseline musculoskeletal ultrasound biomarkers predictive of time-to-flare of arthritis activity following DMARD cessation, including presence or absence of greyscale synovitis/tenosynovitis and erosions.
Genetic biomarkers of DMARD-free remission | At recruitment
  Baseline signature of differential gene expression in peripheral CD4+ T cells predictive of DMARD-free remission at 6 months following DMARD cessation, as measured using RNA sequencing.
Cytokine biomarkers of DMARD-free remission | At recruitment
  Baseline signature of differential cytokine levels in peripheral blood predictive of time-to-flare of arthritis activity, as measured using a multiplex cytokine assay.
Rheumatoid arthritis disease activity | At recruitment and at 1 month, 3 months and 6 months following DMARD cessation
  Measured by Disease Activity Score in 28 joints (DAS28-CRP) score.
Physical disability | At baseline and at 6 months following DMARD cessation
  Measured by Health Assessment Questionnaire Disability Index (HAQ-DI) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: John D Isaacs, PhD MBBS, Principal Investigator — Newcastle University
Locations (1):
- Newcastle NIHR Clinical Research Facility, Royal Victoria Infirmary, Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne & Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No